CLINICAL TRIAL: NCT00148408
Title: Trial of Asthma Patient Education (TAPE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Lung Association Asthma Clinical Research Centers (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: ALAACRC-04
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2006-09

CONDITIONS: Asthma
Keywords: Asthma; Placebo; Education
MeSH Terms: conditions — Asthma | interventions — montelukast; Educational Status

INTERVENTIONS:
Drug: Montelukast
Behavioral: Education

SUMMARY:
The purpose of this research study is to investigate the way that educational approaches and presentation of a drug may affect the response to montelukast and placebo (an inactive medication) in subjects with asthma.

DETAILED DESCRIPTION:
This is a study of the effects of education and drug presentation on efficacy of montelukast and placebo in asthma. This trial will answer the following questions: 1) Is there a true placebo response in asthma that is not due to non-specific factors? 2) Can the placebo effect in asthma be augmented by interventions that increase expectancy of benefit? 3) Can interventions that increase expectancy augment the effect of active treatment? 4) Are placebo effects additive or interactive with treatment effects?

ELIGIBILITY:
Inclusion Criteria:

* age 15 or older
* physician diagnosed asthma
* regular use of prescribed asthma medication over preceding year
* post-bronchodilator FEV1 of at least 75% of predicted
* inadequate asthma control over preceding two months

Exclusion Criteria:

* current or past smoking (greater than 10 pack-years)
* serious asthma exacerbation within previous three months
* regular use of oral corticosteroids
* history of respiratory failure due to asthma
* current use of montelukast or history of adverse reaction to montelukast
* concomitant interfering medical condition
* participation in another clinical trial
* inability or unwillingness to perform study procedures
* pregnancy, lack of effective contraception (when appropriate), lactation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Morning peak expiratory flow

SECONDARY OUTCOMES:
Spirometry
Asthma diaries
Asthma questionnaires (Asthma Control Score, Asthma Symptom Utility Index, Asthma Quality of Life)
Generic health quality of life (SF-36)
Shortness of Breath Questionnaire
Adherence monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Anthonisen, MD, Study Chair — University of Winnipeg
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - National Jewish Hospital, Denver, Colorado
  - Nemour's Childrens Center, Jacksonville, Florida
  - University of Miami (and University of South Florida in Tampa), Miami, Florida
  - Emory University, Atlanta, Georgia
  - Illinois Consortium (Northwestern, Univ. of Chicago, Univ. of Illinois), Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri at Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Long Island Jewish Hospital (and North Shore Hospital), New Hyde Park, New York
  - New York Consortium (New York Univ. and Columbia Univ.), New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Northern New England Consortium (Univ. of Vermont and other locations), Burlington, Vermont

REFERENCES:
- [Derived] Gerald JK, Carr TF, Wei CY, Holbrook JT, Gerald LB. Albuterol Overuse: A Marker of Psychological Distress? J Allergy Clin Immunol Pract. 2015 Nov-Dec;3(6):957-62. doi: 10.1016/j.jaip.2015.06.021. Epub 2015 Sep 1. PMID 26341049
- [Derived] Wise RA, Bartlett SJ, Brown ED, Castro M, Cohen R, Holbrook JT, Irvin CG, Rand CS, Sockrider MM, Sugar EA; American Lung Association Asthma Clinical Research Centers. Randomized trial of the effect of drug presentation on asthma outcomes: the American Lung Association Asthma Clinical Research Centers. J Allergy Clin Immunol. 2009 Sep;124(3):436-44, 444e1-8. doi: 10.1016/j.jaci.2009.05.041. Epub 2009 Jul 25. PMID 19632710
- See also: American Lung Association Asthma Clinical Research Centers — http://www.cctrials.org/alaacrc